CLINICAL TRIAL: NCT05080868
Title: Comparing Epidemiological and Clinical Characteristics of Infantile Hemangioma With Minimal or Arrested Growth (IH-MAG) and Classic Infantile Hemangioma : a Retrospective Study
Brief Title: Infantile Hemangioma With Minimal or Arrested Growth : Epidemiology, Clinical Characteristics and Evolution
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI221
Record Dates: First submitted 2021-03-12; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Hemangioma, Capillary
MeSH Terms: conditions — Hemangioma, Capillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infantile hemangioma with minimal or arrested growth: Epidemiological and clinical characteristics of infantile hemangioma with minimal or arrested growth.
- Classic infantile hemangioma: Epidemiological and clinical characteristics of classic infantile hemangioma.

SUMMARY:
Infantile hemangioma (IH) is the most common vascular tumor of infancy, characterized by its clinical history. Absent at birth or present under the form of a premonitory mark, they display a rapid proliferative phase starting in the first weeks of life. Then, after a plateau phase, they slowly involute. However, a subtype of IH named "abortive", "minimal or arrested growth", "reticular" or "telangiectatic" hemangioma differs from typical IH because it doesn't have a proliferative component, or only a minimal one. This subtype of hemangioma has been recently described and data are lacking regarding its proportion among infantile hemangioma and its differences with "classic" infantile hemangioma. The aim of this study is to estimate the proportion of abortive hemangioma among infantile hemangioma. Also, the investigators aim to compare the clinical characteristics of "classic" infantile hemangiomas and abortive hemangiomas. Lastly, investigators wished to study the evolution of abortive hemangioma.

ELIGIBILITY:
Inclusion Criteria:

* Children between 0 and 18 years old
* Followed in the dermatology department of CHRU de Nancy between January 2014 and December 2020
* Presenting with one or more infantile hemangioma

Exclusion Criteria:

- Those whoes guardian does not want his data to be collected in this study

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: - Children between 0 and 18 years old followed in the dermatology department of CHRU de Nancy between January 2014 and December 2020 presenting with one or more infantile hemangioma
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Proportion of abortive hemangioma among infantile hemangioma | baseline
  Proportion of abortive hemangioma among infantile hemangioma

SECONDARY OUTCOMES:
To compare the epidemiological characteristics between infantile hemangioma and abortive hemangioma : sex | baseline
  Compare sex predominance between infantile hemangioma and abortive hemangioma
To compare the epidemiological characteristics between infantile hemangiomas and abortive hemangiomas : prematurity | baseline
  Compare prematurity rates between infantile hemangiomas and abortive hemangiomas
To compare the epidemiological characteristics between infantile hemangiomas and abortive hemangiomas : birthweight | baseline
  Compare birthweight between infantile hemangiomas and abortive hemangiomas
To compare the clinical characteristics between infantile hemangiomas and abortive hemangiomas : localization | baseline
  Compare localization between infantile hemangiomas and abortive hemangiomas
To compare the clinical characteristics between infantile hemangiomas and abortive hemangiomas : treatment | baseline
  le hemangiomas and abortive hemangiomaCompare treatment between infanti
To compare the clinical characteristics between infantile hemangiomas and abortive hemangiomas : complications | baseline
  Compare complications between infantile hemangiomas and abortive hemangioma
To compare the clinical characteristics between infantile hemangiomas and abortive hemangiomas : size | baseline
  Compare size (focal, extended or segmental) between infantile hemangiomas and abortive hemangioma
To study the evolution of abortive hemangioma : erythematous macule | through study completion, an average of 4 years
  Evaluation of the fading of erythematous macule between the stage of maximal proliferation and the last follow-up
To study the evolution of abortive hemangioma : papules of proliferation | through study completion, an average of 4 years
  Evaluation of the regression of the papules of proliferation between the stage of maximal proliferation and the last follow-up
To study the evolution of abortive hemangioma : telangiectasias | through study completion, an average of 4 years
  Evaluation of the fading of telangiectasias between the stage of maximal proliferation and the last follow-up
To study the evolution of abortive hemangioma : halo of vasoconstriction | through study completion, an average of 4 years
  Evaluation of the fading of the vasoconstricted halo between the stage of maximal proliferation and the last follow-up
To study the evolution of abortive hemangioma : areas of vasoconstriction | through study completion, an average of 4 years
  Evaluation of the fading of vasoconstricted areas between the stage of maximal proliferation and the last follow-up
To study the evolution of abortive hemangioma : dilated veins | through study completion, an average of 4 years
  Evaluation of the fading of dilated veins between the stage of maximal proliferation and the last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: BURSZTEJN Anne-Claire, MD, PhD, Study Director — Central Hospital, Nancy, France
Locations (1):
- CHRU de Nancy, Nancy, Grand Est, France

IPD SHARING:
Plan to Share IPD: No